CLINICAL TRIAL: NCT06993740
Title: The Effect of Dexmedetomidine Administration on the Success of Reconstructive Microsurgery in Cancer Patients: A Study of Glycocalyx Integrity, Inflammatory Response, Thrombosis, Angiogenesis, Oxidative Stress, and Tissue Microcirculation
Brief Title: Effect of Dexmedetomidine on Microsurgery Reconstruction in Cancer Patient
Acronym: DEXFLAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, Gardian Lukman Hakim, Anestesiologist, Dharmais National Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP.04.03/D.XII/5182/2025
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Flap Monitoring; Inflammation; Thrombosis; Oxidative Stress; Glycocalyx; Anesthesia; Surgery; Flap Ischemia; Flap Necrosis; Flap Failure Risk Factors; Microsurgery
Keywords: SOD-1; IL-6; IL-10; VEGF; Syndecan-1; Dexmedetomidine; SDF; PAI-1; Flap Failure; Flap Salvage
MeSH Terms: conditions — Inflammation; Thrombosis | interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the impact of perioperative dexmedetomidine administration on the success of microsurgical reconstruction in cancer patients. The intervention group will receive dexmedetomidine infusion during surgery, while the control group will receive a placebo. The study focuses on assessing surgical outcomes, particularly flap survival, alongside biochemical and histological markers related to endothelial glycocalyx integrity, inflammatory response, thrombosis, angiogenesis, oxidative stress, and microcirculatory function.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial employs a double-blind masking design in which both participants and clinical staff, including surgeons and outcome assessors, are blinded to the treatment allocation. The dexmedetomidine and placebo infusions will be prepared and administered by an independent pharmacist or designated unblinded personnel not involved in patient care or data collection, ensuring unbiased assessment of outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants in this arm will receive a continuous intravenous infusion of placebo (normal saline) administered in the same manner and duration as the dexmedetomidine group-starting after anesthesia induction and continuing for up to 48 hours postoperatively. This control infusion allows comparison of clinical and biochemical outcomes without the influence of dexmedetomidine.
  Interventions: Drug: NaCl 0,9%
- Dexmedetomidine Group (Active Comparator): Participants assigned to this arm will receive a continuous intravenous infusion of dexmedetomidine starting after anesthesia induction and maintained throughout the surgical procedure as well as for up to 48 hours postoperatively. The infusion dose will be titrated to achieve target sedation levels while maintaining stable hemodynamics. This extended administration aims to investigate the effects of dexmedetomidine on endothelial glycocalyx preservation, inflammation modulation, thrombosis prevention, angiogenesis promotion, oxidative stress reduction, and improvement of tissue microcirculation during both intraoperative and early postoperative periods.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: NaCl 0,9% — NaCl 0.9% continuous intravenous infusion during microsurgical reconstruction surgery in cancer patients, started after anesthesia induction and maintained intraoperatively and up to 48 hours postoperatively.
  Other Names: Normal Saline
  Arms: Placebo Group
Drug: Dexmedetomidine — Dexmedetomidine continuous intravenous infusion during microsurgical reconstruction surgery in cancer patients, started after anesthesia induction and maintained intraoperatively and up to 48 hours postoperatively, titrated to maintain target sedation and hemodynamic stability.
  Other Names: Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine Group

SUMMARY:
This double-blinded randomized controlled trial aims to investigate the effect of intraoperative dexmedetomidine administration on early flap viability and microvascular integrity in cancer patients undergoing elective microvascular reconstructive surgery. The primary outcome is clinical flap viability within 48 hours postoperatively, assessed using a standardized scoring system based on flap color, temperature, capillary refill time, and tissue turgor. Secondary outcomes include the evaluation of biomarkers related to endothelial glycocalyx degradation (syndecan-1), oxidative stress (SOD-1), inflammation (IL-6, IL-10), thrombosis (PAI-1), and angiogenesis (VEGF), as well as microcirculatory assessment using Sidestream Dark Field (SDF) imaging. The study is designed to determine whether dexmedetomidine improves early surgical outcomes by modulating pathophysiological processes involved in microvascular flap success.

DETAILED DESCRIPTION:
Microvascular reconstructive surgery is commonly performed in cancer patients following tumor excision to restore both form and function. However, flap failure remains a major postoperative complication, particularly in oncologic patients who are more susceptible to inflammation, endothelial injury, thrombosis, and impaired tissue perfusion. Recent evidence suggests that anesthetic agents may play a role in modulating microvascular and endothelial responses during surgery, providing opportunities to enhance surgical outcomes.

Dexmedetomidine is a selective alpha-2 adrenergic receptor agonist known for its sedative, analgesic, sympatholytic, and anti-inflammatory properties. In addition to its hemodynamic stability profile, dexmedetomidine has demonstrated protective effects on the endothelium and glycocalyx, along with potential benefits in preserving tissue perfusion and reducing inflammatory and thrombotic responses. However, its clinical impact on microvascular flap outcomes in cancer patients undergoing reconstructive surgery has not been well established.

This study is a double-blinded randomized controlled trial involving 60 adult cancer patients (aged 18 to 65 years) undergoing elective microvascular reconstructive surgery. Participants will be randomized into two groups: an intervention group receiving intravenous dexmedetomidine, and a control group receiving normal saline. Both infusions will be prepared in identical syringes to maintain allocation concealment.

The primary outcome of this study is flap viability within the first 48 hours postoperatively, assessed using a standardized clinical scoring system. This scoring incorporates four key parameters: flap color, surface temperature, capillary refill time, and tissue turgor. Each parameter is evaluated to provide an integrated assessment of early microvascular flap function.

The secondary outcomes include exploratory analysis of biological processes related to microvascular integrity and function. These outcomes include the evaluation of biomarkers indicative of endothelial glycocalyx degradation (syndecan-1), oxidative stress (SOD-1), inflammatory activity (IL-6 and IL-10), prothrombotic state (PAI-1), and angiogenesis (VEGF). These markers will be analyzed from plasma and/or flap tissue at defined perioperative time points to better understand the physiological impact of dexmedetomidine.

Furthermore, real-time assessment of tissue microcirculation will be performed using Sidestream Dark Field (SDF) imaging, a non-invasive technique that enables visualization of capillary density and flow quality in the reconstructed flap area. This provides an objective and dynamic measure of tissue-level perfusion and complements the clinical viability scoring.

All patients will undergo general anesthesia induced with fentanyl 2 µg/kg and propofol 1-2 mg/kg. In the intervention group, dexmedetomidine will be administered with a loading dose of 1 µg/kg over 10 minutes, followed by a continuous infusion at 0.4 µg/kg/hour until 48 hours after surgery. The control group will receive a matched volume of normal saline according to the same timeline.

This study is expected to provide new insights into the role of dexmedetomidine in enhancing microvascular outcomes in cancer patients undergoing reconstructive surgery, potentially offering a simple yet impactful strategy to improve flap success and postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 18-65 years) diagnosed with cancer who are scheduled to undergo microsurgical flap reconstruction.
2. Patients within the age range of 18 to 65 years at the time of enrollment.
3. Patients who provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with a history of uncontrolled diabetes mellitus.
2. Patients diagnosed with chronic kidney disease.
3. Patients with known liver failure.
4. Patients receiving corticosteroid therapy prior to surgery.
5. Patients with uncontrolled hypertension.
6. Patients with a history of chemotherapy or radiotherapy prior to surgery.
7. Patients diagnosed with preoperative sepsis.
8. Patients requiring perioperative vasopressor support.
9. Patients with a history of prior surgery in the same operative field.
10. Patients who decline to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Flap Viability Score | 48 hours postoperatively
  Clinical evaluation of flap viability using a standardized scoring system based on four parameters: flap color, surface temperature, capillary refill time, and tissue turgor. Each parameter is scored individually and combined into a composite viability score. The total score reflects the degree of perfusion and tissue viability at 48 hours after microsurgical reconstruction.

SECONDARY OUTCOMES:
Tissue Syndecan-1 Expression | Intraoperative tissue sampling
  Quantitative evaluation of syndecan-1 expression in flap tissue using immunohistochemistry (IHC) to assess endothelial glycocalyx integrity. Image analysis software will be used for objective quantification.
Tissue Superoxide Dismutase 1 (SOD1) Expression | Intraoperative tissue sampling
  Quantitative analysis of SOD1 expression in flap tissue using IHC, serving as a marker of oxidative stress response. Expression will be measured using image-based digital quantification.
Interleukin-6 (IL-6) Level | Baseline (preoperative) and 12 hours postoperatively
  Measurement of systemic IL-6 concentrations using Electrochemiluminescence Immunoassay (ECLIA) as an indicator of systemic inflammatory response.
Interleukin-10 (IL-10) Level | Baseline (preoperative) and 12 hours postoperatively
  Quantification of serum IL-10 levels using Enzyme-Linked Immunosorbent Assay (ELISA), to evaluate anti-inflammatory cytokine response.
Vascular Endothelial Growth Factor (VEGF) Level | Baseline (preoperative) and 12 hours postoperatively
  Assessment of systemic angiogenic activity by measuring VEGF levels in serum using ELISA.
Plasminogen Activator Inhibitor-1 (PAI-1) Level | Baseline (preoperative) and 12 hours postoperatively
  Measurement of PAI-1 levels in serum using ELISA to evaluate the fibrinolytic balance and thrombotic tendency.
Microcirculation Assessment Using Sidestream Dark Field (SDF) Imaging | Immediate postoperative (sublingual site), 12 hours postoperative (flap tissue), and 48 hours postoperative (flap tissue)
  Evaluation of microcirculatory parameters using SDF imaging, including vessel density, perfused vessel density, and flow pattern. Measurements will be conducted at the sublingual site and in the flap tissue at specified time points to assess systemic and local microcirculatory dynamics.

CONTACTS AND LOCATIONS:
Locations (1):
- Dharmais National Cancer Center Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient confidentiality and the limited scope of data use as outlined in the informed consent. The collected data will be used solely for the purposes of this specific clinical study and will not be made publicly available.

REFERENCES:
- [Background] Petersen SM, Greisen G, Hyttel-Sorensen S, Hahn GH. Sidestream dark field images of the microcirculation: intra-observer reliability and correlation between two semi-quantitative methods for determining flow. BMC Med Imaging. 2014 May 6;14:14. doi: 10.1186/1471-2342-14-14. PMID 24885423
- [Background] Atmodiwirjo P, Priambodo PS, Dilogo IH. Pengaruh Titrasi Indocyanine Green terhadap Intensitas Fluoresensi pada Perfusi Flap Bebas dalam Menunjang Tindakan Bedah Mikro Rekonstruksi: Tinjauan terhadap Suhu, TcPCO2, TcPO2, Ekspresi HIF-1α, dan Histopatologi Flap. Universitas Indonesia; 2024.
- [Background] Preidl RHM, Reuss S, Neukam FW, Kesting M, Wehrhan F. Endothelial inflammatory and thrombogenic expression changes in microvascular anastomoses - An immunohistochemical analysis. J Craniomaxillofac Surg. 2021 May;49(5):422-429. doi: 10.1016/j.jcms.2021.02.006. Epub 2021 Feb 12. PMID 33608202
- [Background] Chen Z, Shao DH, Mao ZM, Shi LL, Ma XD, Zhang DP. Effect of dexmedetomidine on blood coagulation in patients undergoing radical gastrectomy under general anesthesia: A prospective, randomized controlled clinical trial. Medicine (Baltimore). 2018 Jul;97(27):e11444. doi: 10.1097/MD.0000000000011444. PMID 29979445
- [Background] Fang M, He J, Ma X, Li W, Lin D. Protective effects of dexmedetomidine on the survival of random flaps. Biomed Pharmacother. 2020 Aug;128:110261. doi: 10.1016/j.biopha.2020.110261. Epub 2020 May 20. PMID 32446114
- [Background] Wijanarko B, Airlangga PS, Fitriati M, Sumartono C, Kriswidyatomo P, Lestari P. Effect of dexmedetomidine administration on malondialdehyde levels in lower extremity surgery using tourniquets. Bali Medical Journal. 2023 May 6;12(2):1459-65.
- [Background] Li B, Li Y, Tian S, Wang H, Wu H, Zhang A, Gao C. Anti-inflammatory Effects of Perioperative Dexmedetomidine Administered as an Adjunct to General Anesthesia: A Meta-analysis. Sci Rep. 2015 Jul 21;5:12342. doi: 10.1038/srep12342. PMID 26196332
- [Background] Hsu TC, Lin CH, Sun FJ, Chen MJ. Postoperative Serum Levels of Interleukin-6 are Affected by Age in Patients with Colorectal Cancer. Int J Gerontol. 2017 Jun;11(2):75-9.
- [Background] Finke JC, Yang J, Bredell M, Fritschen U von, Glocker MO. Plasma Cytokine and Growth Factor Profiling during Free Flap Transplantation. In: Issues in Flap Surgery. InTech; 2018.
- [Background] Lei D, Sha Y, Wen S, Xie S, Liu L, Han C. Dexmedetomidine May Reduce IL-6 Level and the Risk of Postoperative Cognitive Dysfunction in Patients After Surgery: A Meta-Analysis. Dose Response. 2020 Feb 5;18(1):1559325820902345. doi: 10.1177/1559325820902345. eCollection 2020 Jan-Mar. PMID 32076394
- [Background] Yuki K. The immunomodulatory mechanism of dexmedetomidine. Int Immunopharmacol. 2021 Aug;97:107709. doi: 10.1016/j.intimp.2021.107709. Epub 2021 Apr 29. PMID 33933842
- [Background] Abassi Z, Armaly Z, Heyman SN. Glycocalyx Degradation in Ischemia-Reperfusion Injury. Am J Pathol. 2020 Apr;190(4):752-767. doi: 10.1016/j.ajpath.2019.08.019. Epub 2020 Feb 6. PMID 32035883
- [Background] Pillinger NL, Kam P. Endothelial glycocalyx: basic science and clinical implications. Anaesth Intensive Care. 2017 May;45(3):295-307. doi: 10.1177/0310057X1704500305. PMID 28486888
- [Background] Pang CY, Neligan PC. Flap Pathophysiology and Pharmacology. In: Gurtner GC, Neligan PC, editors. Plastic Surgery, Volume 1: Principles. Fourth Ed. Canada: Elsevier Inc.; 2018. p. 433-443.e7.
- [Background] Sigaux N, Philouze P, Boucher F, Jacquemart M, Frobert P, Breton P. Efficacy of the postoperative management after microsurgical free tissue transfer. J Stomatol Oral Maxillofac Surg. 2017 Jun;118(3):173-177. doi: 10.1016/j.jormas.2017.03.007. Epub 2017 Apr 5. PMID 28391079
- [Background] Han M, Ochoa E, Zhu B, Park AM, Heaton CM, Seth R, Knott PD. Risk Factors for and Cost Implications of Free Flap Take-backs: A Single Institution Review. Laryngoscope. 2021 Jun;131(6):E1821-E1829. doi: 10.1002/lary.29382. Epub 2021 Jan 13. PMID 33438765
- [Background] Pu LLQ, Song P. Reoperative Microsurgical Free Flap Surgery: Lessons Learned. Ann Plast Surg. 2023 May 1;90(5S Suppl 2):S187-S194. doi: 10.1097/SAP.0000000000003370. Epub 2023 Jan 18. PMID 36752558
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Riskesdas. Hasil Utama Riskesdas 2018. Kementrian Kesehatan Republik Indonesia. 2018.